CLINICAL TRIAL: NCT03381976
Title: Effects of Different Frequency Low-volume Resistance Training on Body Fat in Obese Older: A Randomized Controlled Trial
Brief Title: Body Fat and Frequency of Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Crisieli Maria Tomeleri, Doctor, Universidade Estadual de Londrina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UEL09167-2/2015
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 2X/week (G2X) (Active Comparator): This group performed resistance training twice a week (Tuesdays and Thursdays)
  Interventions: Other: Intervention 2X/week (G2X)
- Intervention 3X/week (G3X) (Active Comparator): This group performed resistance training three sessions a week (Mondays, Wednesdays, and Fridays).
  Interventions: Other: Intervention 3X/week (G3X)
- Control group (GC) (No Intervention): This group did not perform any type of organized physical exercise during the study period.

INTERVENTIONS:
Other: Intervention 2X/week (G2X) — Participants performed resistance training (RT) composed of eight exercises performed for one set of 10-15 repetition maximum (RM). The rest interval between exercises was 2-3 min. Participants were instructed to control the speed of movement in the ratio of 1:2 for concentric and eccentric muscle actions, respectively. The progression of training loads in each exercise occurred, when a participant completed 15 repetitions in two consecutive sessions, with increases of 2-5% in exercises for the upper limbs, and 5-10% in exercises for the lower limbs. At the end of each session, one static stretching exercise at the point of discomfort for 15 seconds was performed for all major muscle groups for a total of exercises. Participants were asked not to perform any other type of organized physical exercise during the entire study period.
  Arms: Intervention 2X/week (G2X)
Other: Intervention 3X/week (G3X) — Participants performed resistance training (RT) composed of eight exercises performed for one set of 10-15 repetition maximum (RM). The rest interval between exercises was 2-3 min. Participants were instructed to control the speed of movement in the ratio of 1:2 for concentric and eccentric muscle actions, respectively. The progression of training loads in each exercise occurred, when a participant completed 15 repetitions in two consecutive sessions, with increases of 2-5% in exercises for the upper limbs, and 5-10% in exercises for the lower limbs. At the end of each session, one static stretching exercise at the point of discomfort for 15 seconds was performed for all major muscle groups for a total of exercises. Participants were asked not to perform any other type of organized physical exercise during the entire study period.
  Arms: Intervention 3X/week (G3X)

SUMMARY:
This study compared different frequency low-volume resistance training (RT) on total, android, gynoid and trunk body fat in obese older women

DETAILED DESCRIPTION:
The aim of this study was to compare the effect of resistance training with different frequencies on total, android, gynoid and trunk body fat in obese older women. Recruitment was carried out through newspaper and radio advertisements, and home delivery flyers in residential neighborhoods. All participants completed health history and physical activity questionnaires, and met the following inclusion criteria: 60 years of age or older, relative body fat ≥ 32 assessed by whole body dual-energy X-ray absorptiometry (DXA), physically independent, free from cardiac or orthopedic dysfunction that would have precluded them from performing the tests or the training program associated with the study, not receiving hormonal replacement therapy, and not performing physical exercise more than once a week in the six months preceding the beginning of the investigation.Written informed consent was obtained from all participants after a detailed description of study procedures was provided. This study was conducted in accordance with the Declaration of Helsinki and approved by the local Ethics Research Committee, and was carried out over a period of 16 weeks, with 12 weeks dedicated to the resistance training program, and 4 weeks directed to testing. Anthropometric, body composition, and dietary intake measurements were performed during weeks 1-2, and 15-16. A supervised progressive resistance training was performed between weeks 3-14. The control group did not perform any type of organized physical exercise during the study period. Supervised resistance training was performed during the 12 weeks of training. All participants were individually supervised by physical education professionals throughout each training session to ensure that the study's training protocol was followed and to ensure subject safety. The group 2X performed the program twice a week (Tuesdays and Thursdays), while group 3X performed three sessions a week (Mondays, Wednesdays, and Fridays). The progression of training loads in each exercise occurred, when a participant completed 15 repetitions in two consecutive sessions, with increases of 2-5% in exercises for the upper limbs, and 5-10% in exercises for the lower limbs. At the end of each session, one static stretching exercise at the point of discomfort for 15 seconds was performed for all major muscle groups for a total of exercises. Participants were asked not to perform any other type of organized physical exercise during the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older;
* relative body fat ≥ 32 assessed by whole body dual-energy X-ray absorptiometry (DXA);
* physically independent;
* free from cardiac or orthopedic dysfunction that would have precluded them from performing the tests or the training program associated with the study;
* not receiving hormonal replacement therapy;
* not performing physical exercise more than once a week in the six months preceding the beginning of the investigation.

Exclusion Criteria:

• All subjects not participating in 85% of the total sessions of training or withdrawl

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2015-07-24 (Actual)

PRIMARY OUTCOMES:
Change in body composition | baseline and 12 weeks
  Whole-body dual-energy X-ray absorptiometry (DXA) scans (Lunar Prodigy, model NRL 41990, GE Lunar, Madison, WI) were used to assess total body fat, trunk fat, gynoid fat and android fat. Prior to scanning, participants were instructed to remove all objects containing metal. Scans were performed with the subjects lying in the supine position along the table's longitudinal centerline axis. Feet were taped together at the toes to immobilize the legs while the hands were maintained in a pronated position within the scanning region. Both calibration and analysis were carried out by a skilled laboratory technician. Equipment calibration followed the manufacturer's recommendations. The software generated standard lines that set apart the limbs from the trunk and head. These lines were adjusted by the same technician using specific anatomical points determined by the manufacturer. The results are presented in kilograms (kg)
Change in fat z-score | baseline and 12 weeks
  A composite z-score, was calculated using the following formula: (total body fat z-score) + (gynoid body fat z-score) + (android fat z-score) / 3. Z-scores were obtained from the DXA using standard software.

SECONDARY OUTCOMES:
Changes in Anthropometry Parameters | baseline and 12 weeks
  Body mass was measured to the nearest 0.1 kg using a calibrated electronic scale (Balmak, Laboratory Equipment Labstore, Curitiba, Paraná, Brazil), with the participants wearing light workout clothing and no shoes. Height was measured with a stadiometer attached to the scale to the nearest 0.1 cm, with subjects standing without shoes. These parameter will be combined to report body mass index that will be calculate as body mass in kilograms divided by the square of height in meters.
Changes in Dietary intake | baseline and 12 weeks
  Participants were instructed by a dietitian to complete a food record on three nonconsecutive days (two week days and one weekend day) pre- and post-intervention. Participants were given specific instructions regarding the recording of portion sizes and quantities to identify all food and fluid intake, in addition to viewing food models in order to enhance precision. The amount of protein, carbohydrate, and lipid were calculated using nutrition analysis software (Avanutri Processor Nutrition Software, Rio de Janeiro, Brazil; Version 3.1.4). The sum of the three macronutrients will be presented by total energy intake which will be expressed per kcal/kg per day.
Changes in Total Strength | baseline and 12 weeks
  Maximal dynamic strength was evaluated using the one repetition maximum (1RM) test assessed in the chest press, knee extension, and preacher curl exercises, performed in this exact order. Testing for each exercise was preceded by a warmup set (6-10 repetitions), with approximately 50% of the estimated load used in the first attempt of the 1RM. This warmup was also used to familiarize the subjects with the testing equipment and lifting technique. The testing procedure was initiated 2 minutes after the warm-up. The subjects were instructed to try to accomplish two repetitions with the imposed load and were given three attempts in both exercises. The rest period was 3 to 5 min between each attempt, and 5 min between exercises. The 1RM was recorded as the final load lifted in which the subject was able to complete only one single maximal execution. Total strength was determined by the sum of the 3 exercises, expressed in kg.

IPD SHARING:
Plan to Share IPD: No